CLINICAL TRIAL: NCT01203930
Title: A Phase 2 Single Arm Study to Investigate the Safety and Clinical Activity of Idelalisib Alone and in Combination With Rituximab in Elderly Subjects With Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: A Study of Idelalisib and Rituximab in Elderly Patients With Untreated CLL or SLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-08
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: CLL; SLL; GS-1101; CAL-101; Phosphatidylinositol 3-kinase (PI3K); Rituximab; Rituxan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental): This arm consists of 2 cohorts. Participants in Cohort 1 will receive idelalisib for up to twelve 28-day cycles (or development of unacceptable toxicity) plus rituximab (8 doses through the end of Cycle 2). Upon completion of twelve 28-cycles, participants are eligible to remain on idelalisib in a continuation protocol. Participants in Cohort 2 will receive idelalisib until disease progression or development of unacceptable toxicity.
  Interventions: Drug: Idelalisib; Drug: Rituximab

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg tablets administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101
Drug: Rituximab — Rituximab 375 mg/m^2 administered intravenously once weekly x 8 weeks
  Other Names: Rituxan

SUMMARY:
This study is to evaluate the safety and clinical activity of idelalisib alone and in combination with rituximab in patients with CLL or SLL.

This Phase 2 study will be the first time that idelalisib is administered to previously untreated patients with hematologic malignancies. Idelalisib has demonstrated clinical activity as a single agent in relapsed or refractory CLL and SLL with acceptable toxicity, which supports its evaluation in previously untreated patients. The study population is limited to patients over 65 years of age because younger patients are generally appropriate for standard immunochemotherapy regimens that are highly active. Since the mechanism of action of idelalisib is distinct from rituximab, it is hypothesized that the combination will be more active than either agent alone. This study will establish initial safety and clinical activity of idelalisib in combination with rituximab in patients with CLL or SLL. Cohort 2 of this study will establish safety and clinical activity of idelalisib alone in subjects with untreated CLL or SLL.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed CLL or SLL.
* Age ≥ 65
* Presence of measurable lymphadenopathy (defined as the presence of ≥1 nodal lesion that measures ≥ 1.5 cm in the longest diameter (LD) and ≥ 1.0 cm in the longest perpendicular diameter (LPD) as assessed by physical exam, computed tomography (CT) or magnetic resonance imaging (MRI)).
* CLL - Binet Stage C or Rai Stage III or IV or has active disease defined by meeting at least one of the following criteria:

  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
  * Massive (ie, > 6 cm below the left costal margin) or progressive or symptomatic splenomegaly
  * Massive nodes (ie, > 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy
  * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or lymphocyte doubling time of less than 6 months
  * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids or other standard therapy
  * At least one of the following disease-related symptoms:

    * Unintentional weight loss ≥ 10% within the previous 6 months
    * Significant fatigue
    * Fevers > 100.4 F for ≥ 2 weeks without other evidence of infection
    * Night sweats for ≥ 1 month without evidence of infection
* SLL - has active disease as defined above for CLL, except the lymphocytosis criterion does not apply
* World Health Organization (WHO) Performance Status of ≤ 2
* For men of child-bearing potential, willing to use adequate methods of contraception for the entire duration of the study
* Able to provide written informed consent

Key Exclusion Criteria:

* Prior therapy for CLL or SLL, except corticosteroids for symptom relief
* Treatment with a short course of corticosteroids for symptom relief within 1-week prior to Visit 1
* Known active central nervous system involvement of the malignancy
* Ongoing active, serious infection requiring systemic therapy. Patients may be receiving prophylactic antibiotics and antiviral therapy at the discretion of the treating physician.
* Serum creatinine ≥ 2.0 mg/dL
* Serum bilirubin ≥ 2 mg/dL (unless due to Gilbert's syndrome) or serum transaminases (ie, aspartate aminotransferase (AST), alanine aminotransferase (ALT)) ≥ 2 x upper limit of normal
* Positive test for human immunodeficiency virus (HIV) antibodies
* Active hepatitis B or C (confirmed by ribonucleic acid (RNA) test). Patients with serologic evidence of prior exposure are eligible.
* History of a non-CLL malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to study entry, other adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 5 years.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - University of California, San Diego, Moores Cancer Center, La Jolla, California
  - Stanford University School of Medicine, Stanford, California
  - Columbia University - Herbert Irving Pavilion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The Universtity of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] O'Brien SM, Lamanna N, Kipps TJ, Flinn I, Zelenetz AD, Burger JA, Keating M, Mitra S, Holes L, Yu AS, Johnson DM, Miller LL, Kim Y, Dansey RD, Dubowy RL, Coutre SE. A phase 2 study of idelalisib plus rituximab in treatment-naive older patients with chronic lymphocytic leukemia. Blood. 2015 Dec 17;126(25):2686-94. doi: 10.1182/blood-2015-03-630947. Epub 2015 Oct 15. PMID 26472751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 28 September 2010. The last study visit occurred on 07 June 2016.
Pre-assignment Details: 113 participants were screened.
Groups:
- Idelalisib+Rituximab (Cohort 1): Idelalisib 150 mg capsules or tablets administered orally twice daily of each 28-day cycle for 12 cycles + rituximab 375 mg/m^2 administered intravenously weekly for 8 doses
- Idelalisib (Cohort 2): Idelalisib 150 mg capsules or tablets administered orally twice daily of each 28-day cycle until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Started | 64 | 41
Completed | 43 (43 participants completed 12 cycles and were then eligible to enroll in the extension study (101-99)) | 0
Not Completed | 21 | 41
Not completed — Disease Progression | 0 | 4
Not completed — Death | 3 | 1
Not completed — Withdrew Consent | 1 | 10
Not completed — Investigator Request | 0 | 8
Not completed — Study Terminated by Sponsor | 0 | 12
Not completed — Poor tolerance of study drug | 0 | 1
Not completed — Adverse Event | 17 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Set: participants who received at least 1 dose of idelalisib.
Groups:
- Idelalisib+Rituximab (Cohort 1): Idelalisib 150 mg capsules or tablets administered orally twice daily of each 28-day cycle for 12 cycles + rituximab 375 mg/m^2 administered intravenously weekly for 8 doses. Participants who completed 12 cycles of idelalisib were eligible to continue treatment on an extension study (101-99).
- Total: Total of all reporting groups
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2) | Total
Number analyzed (Participants) | 64 | 41 | 105
Age, Customized [Number; unit: participants]
  < 70 Years | 29 | 14 | 43
  ≥ 70 Years | 35 | 27 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 40 | 32 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 64 | 40 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 61 | 40 | 101
  Black or African American | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was assessed based on standardized International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria as specifically modified for this study to reflect current recommendations which consider the mechanism of action of idelalisib and similar drugs, and was defined as the proportion of participants achieving a complete response (CR) or partial response (PR) as assessed by the investigator. Based on the CLL response definition in the protocol (modified Hallek 2008), the parameters of lymphadenopathy, liver and/or spleen size, constitutional symptoms, polymorphonuclear leukocytes, circulating clonal B-lymphocytes, platelet count, hemoglobin, and marrow were assessed.
  * CR: meeting all defined criteria
  * PR: meeting at least 2 of the criteria of circulating lymphocytes, lymphadenopathy, liver, spleen, or bone marrow (or only lymphadenopathy if liver and spleen normal at baseline) and at least 1 of the criteria for polymorphonuclear leukocytes, platelet count, or hemoglobin.
Time Frame: Up to 28 Months
Population: Intent-to-treat (ITT) Analysis Set: participants who received at least 1 dose of idelalisib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 64 | 41
percentage of participants | 96.9 [89.2 to 99.6] | 87.8 [73.8 to 95.9]

2. Secondary Outcome: Overall Safety of Idelalisib
Description: The overall safety of idelalisib was assessed as the percentage of participants experiencing treatment-emergent adverse events (AEs; Serious AEs, Grade ≥ 3 AEs, AEs related to idelalisib, and AEs leading to discontinuation of idelalisib).
Time Frame: Up to 28 Months
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 64 | 41
percentage of participants
  Any AE | 100.0 | 100.0
  Serious AE | 48.4 | 68.3
  Grade ≥ 3 AE | 76.6 | 85.4
  AE related to idelalisib | 81.3 | 97.6
  AE leading to permanent drug discontinuation | 28.1 | 56.1

3. Secondary Outcome: Lymphadenopathy Response Rate
Description: Lymphadenopathy response rate was defined as the percentage of participants with a ≥ 50% reduction from baseline in the sum of the perpendicular diameters of all measurable lesions while receiving study therapy.
Time Frame: Baseline and up to 28 Months
Population: Participants in the ITT Analysis Set with baseline measurable lymph nodes were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 50 | 38
percentage of participants | 98.0 [89.4 to 99.9] | 86.8 [71.9 to 95.6]

4. Secondary Outcome: Percent Change From Baseline in the Sum of the Product of the Greatest Perpendicular Diameters (SPD) of All Measurable Lesions
Time Frame: Baseline; Weeks 8, 16, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: percent change
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 50 | 38
percent change
  % Change at Wk 8: number analyzed (Participants) | 47 | 20
  % Change at Wk 8 | -100.0 [-100.0 to -8.3] | -69.8 [-100.0 to 0.0]
  % Change at Wk 16: number analyzed (Participants) | 40 | 16
  % Change at Wk 16 | -100.0 [-100.0 to -69.2] | -74.5 [-100.0 to 0.0]
  % Change at Wk 24: number analyzed (Participants) | 43 | 26
  % Change at Wk 24 | -100.0 [-100.0 to -50.0] | -76.0 [-100.0 to 0.0]
  % Change at Wk 36: number analyzed (Participants) | 30 | 10
  % Change at Wk 36 | -100.0 [-100.0 to -66.7] | -77.5 [-100.0 to 0.0]
  % Change at Wk 48: number analyzed (Participants) | 33 | 18
  % Change at Wk 48 | -100.0 [-100.0 to -50.0] | -73.9 [-98.3 to 44.4]
  % Change at Wk 60: number analyzed (Participants) | 0 | 9
  % Change at Wk 60 |  | -69.7 [-93.3 to -56.7]
  % Change at Wk 72: number analyzed (Participants) | 0 | 5
  % Change at Wk 72 |  | -78.0 [-85.5 to -68.8]
  % Change at Wk 84: number analyzed (Participants) | 0 | 3
  % Change at Wk 84 |  | -80.0 [-91.2 to -68.1]
  % Change at Wk 96: number analyzed (Participants) | 0 | 2
  % Change at Wk 96 |  | -81.3 [-100.0 to -62.5]
  % Change at Wk 108: number analyzed (Participants) | 0 | 1
  % Change at Wk 108 |  | -78.1 [-78.1 to -78.1]
  % Change at Wk 120: number analyzed (Participants) | 0 | 1
  % Change at Wk 120 |  | -71.9 [-71.9 to -71.9]
  Best % Change | -100.0 [-100.0 to -40.0] | -81.1 [-100.0 to 0.0]

5. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of disease progression or death from any cause.
Time Frame: Up to 28 Months
Population: Participants in the ITT Analysis Set who achieved complete or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 62 | 35
months | NA [NA to NA] — NA: Not reached | 14.8 [10.0 to NA] — NA: Not reached

6. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from the first dose date of drug to the earlier of the first documentation of definitive disease progression or death from any cause.
  Progression was defined using the Standardized IWCLL criteria as specifically modified for this study to consider the mechanism of action of idelalisib and similar drugs. The occurrence of any of the following events indicated progression:
  1. Evidence of any new disease
  2. Evidence of worsening of index lesions, spleen or liver, or non-index disease
  3. Decrease in platelet count or hemoglobin that is attributable to CLL and is confirmed by bone marrow biopsy
Time Frame: Up to 28 Months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 64 | 41
months | NA [NA to NA] — Not reached | 26.2 [14.0 to NA] — Not reached

7. Secondary Outcome: Idelalisib Plasma Concentrations (Cohort 1)
Time Frame: Predose and 1.5 hours postdose at Weeks 0, 4, and 24
Population: Pharmacokinetic (PK) Analysis Set: participants in the ITT Analysis Set from Cohort 1 who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Idelalisib+Rituximab (Cohort 1)
Number analyzed (Participants) | 64
ng/mL
  Week 0 predose | 0.0 [0.0 to 0.0]
  Week 0 postdose: number analyzed (Participants) | 63
  Week 0 postdose | 1710.0 [1060.0 to 2660.0]
  Week 4 predose: number analyzed (Participants) | 57
  Week 4 predose | 305.0 [189.0 to 606.0]
  Week 4 postdose: number analyzed (Participants) | 52
  Week 4 postdose | 1720.0 [1090.0 to 2500.0]
  Week 24 predose: number analyzed (Participants) | 44
  Week 24 predose | 256.5 [173.5 to 625.5]
  Week 24 postdose: number analyzed (Participants) | 45
  Week 24 postdose | 1460.0 [925.0 to 2010.0]

8. Secondary Outcome: Idelalisib Plasma Concentrations (Cohort 2)
Time Frame: Predose and 1.5 hours postdose at Weeks 0 and 4 and predose at Weeks 8 and 20
Population: PK Analysis Set: participants in the ITT Analysis Set from Cohort 2 who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Idelalisib (Cohort 2)
Number analyzed (Participants) | 40
ng/mL
  Week 0 predose: number analyzed (Participants) | 38
  Week 0 predose | 0.0 [0.0 to 0.0]
  Week 0 postdose | 2190.0 [1575.0 to 2920.0]
  Week 4 predose: number analyzed (Participants) | 30
  Week 4 predose | 293.0 [228.0 to 549.0]
  Week 4 postdose: number analyzed (Participants) | 31
  Week 4 postdose | 2120.0 [1850.0 to 2590.0]
  Week 8 predose: number analyzed (Participants) | 27
  Week 8 predose | 453.0 [207.0 to 904.0]
  Week 20 predose: number analyzed (Participants) | 20
  Week 20 predose | 590.0 [317.0 to 971.5]

9. Secondary Outcome: Changes in Potential Pharmacodynamic Markers of Drug Activity in Plasma and Whole Blood
Description: Changes in potential pharmacodynamic markers of drug activity will include assessments of chemokine and cytokine concentrations, effects on the activity of PI3K and related pathways, and effect on cell migration and other functional outcomes. This endpoint will be assessed at the following time points:
  * Idelalisib+Rituximab (Cohort 1): Predose and 1.5 hour postdose on Day 1 and predose on Days 15, 29, 57, 113, and 169
  * Idelalisib (Cohort 2): Predose on Days 1, 29, 57, 141
Time Frame: Up to 169 days
Population: The collection of plasma samples for pharmacodynamic (PD) analysis in this study was planned prior to the availability of results from an identical PD analysis in another idelalisib study with a larger sample size (n = 176 unique subjects with 2085 longitudinal plasma samples). Therefore, PD analysis was not performed in this study (n = 41).
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the interval from the start of study treatment to death from any cause.
Time Frame: Up to 28 Months
Population: Overall survival analysis was not performed because the follow-up period was insufficient to capture enough events.
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 Months
Description: Adverse events were coded according to MedDRA Version 15.1 for Cohort 1 and MedDRA Version 19.0 for Cohort 2.
Arm/Group | Idelalisib+Rituximab (Cohort 1) | Idelalisib (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 31/64 | 28/41
Other Adverse Events (participants affected / at risk) | 63/64 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Rituximab (Cohort 1) (N=64) | Idelalisib (Cohort 2) (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Cellulitis (Infections and infestations) | 1 | 2
Clostridial infection (Infections and infestations) | 1 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 5
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Rituximab (Cohort 1) (N=64) | Idelalisib (Cohort 2) (N=41)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Neutropenia (Blood and lymphatic system disorders) | 3 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 10
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Colitis (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 11 | 12
Diarrhoea (Gastrointestinal disorders) | 31 | 27
Dry mouth (Gastrointestinal disorders) | 1 | 4
Flatulence (Gastrointestinal disorders) | 4 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 24 | 14
Stomatitis (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 14 | 7
Asthenia (General disorders) | 7 | 0
Chest discomfort (General disorders) | 4 | 0
Chills (General disorders) | 23 | 6
Fatigue (General disorders) | 20 | 13
Influenza like illness (General disorders) | 8 | 1
Malaise (General disorders) | 6 | 1
Oedema (General disorders) | 4 | 2
Oedema peripheral (General disorders) | 8 | 10
Peripheral swelling (General disorders) | 0 | 3
Pyrexia (General disorders) | 26 | 13
Candida infection (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 7 | 4
Sinusitis (Infections and infestations) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Urinary tract infection (Infections and infestations) | 9 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 0
Alanine aminotransferase increased (Investigations) | 18 | 11
Aspartate aminotransferase increased (Investigations) | 17 | 10
Blood alkaline phosphatase increased (Investigations) | 2 | 3
Liver function test abnormal (Investigations) | 6 | 0
Neutrophil count decreased (Investigations) | 2 | 3
Transaminases increased (Investigations) | 9 | 0
Weight decreased (Investigations) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 7 | 1
Dysgeusia (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 15 | 5
Anxiety (Psychiatric disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 13 | 2
Renal failure acute (Renal and urinary disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 10 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 5
Rash (Skin and subcutaneous tissue disorders) | 24 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 7
Flushing (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 3 | 3
Hypotension (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years